CLINICAL TRIAL: NCT07387939
Title: Anterior Cruciate Ligament Reconstruction in Patients Aged 50 Years and Older
Brief Title: ACL Reconstruction in Patients Aged 50 Years and Older
Acronym: LCA Over 50
Status: Active, not recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: LCA Over 50
Record Dates: First submitted 2026-01-08; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: ACL Injury
Keywords: knee; anterior cruciate ligament; ACL reconstruction; elderly patients
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Over 50: ACL reconstructed patients over 50 years of age
- ACl under 40: ACL reconstructed patients under 40 years of age

SUMMARY:
Anterior cruciate ligament (ACL) injury is one of the most common knee ligament injuries in athletes, and surgical ACL reconstruction is the treatment of choice to allow patients to return to sports and recreational activities. Surgical treatment restores joint kinematics, reduces the risk of subsequent injuries, and reduces the degenerative progression of the joint. With the increasing average age, life expectancy, and physical activity levels of the population over 50, ACL injuries are also becoming more frequent in this group. Traditionally, the treatment of choice for patients over 50 has been conservative, based on muscle-strengthening exercises and rescheduling of sports activity with lifestyle modifications to accommodate the joint deficit. Furthermore, some authors have demonstrated that ACL reconstruction in older patients can lead to a higher rate of complications such as stiffness, arthrofibrosis, infections, wound healing problems, or thromboembolic risks, as well as the fact that the presence of concomitant early degenerative osteoarthritis can prevent a satisfactory outcome. Furthermore, studies have shown that nonsurgical treatment may be the most cost-effective strategy in middle-aged patients with moderate activity levels. Currently, there is no consensus regarding the appropriateness of ACL reconstruction in patients over 50, as it is unclear whether there may be greater risks or whether the procedure may lead to more postoperative complications compared to younger patients.

However, several studies have shown that in a middle-aged population with ACL deficiency, selected and motivated patients can experience significant recovery of joint function and stability after surgical reconstruction, with a satisfactory return to sports and recreational activities. There is now growing evidence that surgical treatment can offer favorable outcomes in patients over 50 in terms of knee stability and patient satisfaction, with results similar to those observed in a younger patient population.

General Objective:

The purpose of this study is to evaluate subjective and objective functional outcomes in patients over 50 undergoing ACL reconstruction, comparing them with a population under 40.

The study's hypothesis is that ACL reconstruction surgery in patients over 50 will yield satisfactory clinical results, comparable to those in patients under 40.

Primary Objective:

The purpose of this study is to evaluate subjective and objective functional outcomes in patients over 50 undergoing ACL reconstruction at least two years after surgery.

Secondary Objectives:

Comparison of results with a population under 40.

Patients to be Enrolled:

The minimum sample size was estimated using subjective IKDC assessed at various time points after surgery in a group of patients over 50 years of age as the primary endpoint. The calculation was performed in G*Power (v3.1.9.7) assuming an α error of 0.05, a power (1-β error) of 0.80, and an effect size of 0.625 (1). The minimum estimated sample size is 23 patients. Taking into account any dropouts, an additional 20% of patients will be considered, for a total of 28 patients. To evaluate the effectiveness of the intervention in patients over 50 years of age, subjective functional outcomes will be compared with those of an equal population under 40 years of age (n=28). Therefore, the study requires the enrollment of 56 total patients, 28 per group. A total of 56 patients were divided into the two groups described in the study.

Inclusion Criteria:

* Patients who underwent ACL reconstruction surgery from 2016 to 2021 at our Institute
* Patients who were older than 50 or younger than 40 years of age at the time of surgery
* Signed informed consent and agreed to participate in all study procedures

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will not be enrolled in the study:

* Failure to provide informed consent
* Patients undergoing combined anterior and posterior cruciate ligament reconstruction procedures, patients undergoing combined anterior cruciate ligament reconstruction and prosthetic surgery

Patients enrolled in the study, after signing the informed consent form, will be contacted again to undergo routine assessment procedures, International Knee Documentation Committee (IKDC) score, ACL-RSI (Anterior Cruciate Ligament-Return to Sport after Injury) scale and Tegner activity scale, physical examination including ROM, stability tests such as Lachman and anterior drawer. Demographic variables (i.e., age, sex, body mass index) and surgical data will be collected by an independent researcher.

Translational relevance:

With increasing life expectancy and patient functional needs, and a projected doubling of the middle-aged population by 2050, this study aims to evaluate the effectiveness of ACL reconstruction surgery in subjects over 50 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent ACL reconstruction surgery from 2016 to 2021 at our institution
* Patients who were older than 50 or younger than 40 years of age at the time of surgery
* Signed informed consent and agreed to participate in all study procedures

Exclusion Criteria:

* Non-acceptance of informed consent
* Patients undergoing combined anterior and posterior cruciate ligament reconstruction procedures, patients undergoing combined anterior cruciate ligament reconstruction and prosthetic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent ACl reconstruction
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) subjective form | Through study completion, an average of 2 years
  The International Knee Documentation Committee (IKDC) Subjective Knee Form is a 18-item patient-reported outcome measure used to assess knee symptoms, function, and sports activity, ranging from 0 to 100 (higher is better).

SECONDARY OUTCOMES:
ACL-RSI (Anterior Cruciate Ligament-Return to Sport after Injury) scale | Through study completion, an average of 2 years
  The Anterior Cruciate Ligament-Return to Sport after Injury (ACL-RSI) scale was created to evaluate psychological readiness with regard to Return-to-Sport. It includes 12 items about confidence and fear relative to performance, reinjury, and returning to pre-injury sport participation. It ranges from 0 to 100, where higher scores signify greater confidence, lower fear, and better emotional readiness
Tegner activity level | Through study completion, an average of 2 years
  Tegner Activity Scale (TAS) is a self-administered patient-reported measure that describes the level of work- and sports-based activity in which a patient can engage, ranging from 0 to 10 (higher is better), from Level 0 (Sick leave or disability pension because of knee problems) to Level 10 - Competitive sports: soccer, football, rugby (national or international elite)

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panisset JC, Gonzalez JF, de Lavigne C, Ode Q, Dejour D, Ehlinger M, Fayard JM, Lustig S; French Arthroscopic Society. ACL reconstruction in over-50 year-olds: Comparative study between prospective series of over-50 year-old and under-40 year-old patients. Orthop Traumatol Surg Res. 2019 Dec;105(8S):S259-S265. doi: 10.1016/j.otsr.2019.09.009. Epub 2019 Oct 21. PMID 31648996
- [Background] Figueroa D, Figueroa F, Calvo R, Vaisman A, Espinoza G, Gili F. Anterior cruciate ligament reconstruction in patients over 50 years of age. Knee. 2014 Dec;21(6):1166-8. doi: 10.1016/j.knee.2014.08.003. Epub 2014 Aug 28. PMID 25174853
- [Background] Ehlinger M, Panisset JC, Dejour D, Gonzalez JF, Paihle R, Favreau H, Ollivier M, Lustig S; Francophone Arthroscopy Society (SFA). Anterior cruciate ligament reconstruction in the over-50s. A prospective comparative study between surgical and functional treatment. Orthop Traumatol Surg Res. 2021 Dec;107(8S):103039. doi: 10.1016/j.otsr.2021.103039. Epub 2021 Aug 8. PMID 34375770
- [Background] Salesky MA, Oeding JF, Zhang AL, Ma CB, Feeley BT, Lansdown DA. Patients Aged 50 Years and Older Have Greater Complication Rates After Anterior Cruciate Ligament Reconstruction: A Large Database Study. Arthrosc Sports Med Rehabil. 2021 Oct 9;3(6):e1827-e1834. doi: 10.1016/j.asmr.2021.08.010. eCollection 2021 Dec. PMID 34977637
- [Background] D'Ambrosi R, Giorgino R, Corona K, Jaykumar T, Mariani I, Ursino N, Mangiavini L, Vaishya R. Hamstring tendon autografts and allografts show comparable clinical outcomes and knee stability after anterior cruciate ligament reconstruction in patients over fifty years old with no signs of osteoarthritis progression. Int Orthop. 2022 Sep;46(9):2029-2039. doi: 10.1007/s00264-022-05465-3. Epub 2022 Jun 8. PMID 35672579